CLINICAL TRIAL: NCT03972345
Title: A Non-interventional, Prospective Study in Germany to Investigate the Influence of Adherence to Growth Hormone Therapy (GHT) With Norditropin® on Near Final Height in a Patient Population With Isolated Growth Hormone Deficiency (GHD) and Born Small for Gestational Age (SGA)
Brief Title: Influence of Adherence to Growth Hormone Therapy (GHT) With Norditropin® on Near Final Height in Patients With Growth Hormone Deficiency (GHD) and Born Small for Gestational Age (SGA)
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GH-4488; U1111-1217-5835 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-05-31; First posted 2019-06-03 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Growth Hormone Deficiency in Children; Born Small for Gestational Age

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paediatric patients with iGHD or SGA: Children with one of the following confirmed diagnoses: isolated growth hormone deficiency (iGHD) or small for gestational age (SGA)
  Interventions: Drug: Norditropin® FlexPro®

INTERVENTIONS:
Drug: Norditropin® FlexPro® — Patients will be treated with commercially available Norditropin® FlexPro® according to routine clinical practice at the discretion of the treating physician. The decision to initiate treatment with commercially available Norditropin® FlexPro® has been made by the treating physician and the patient's parents/legal guardian before and independently of the decision to include the patient in this study.

SUMMARY:
Participants are free to decide if they want to take part in this study or not. The study will be conducted to collect information about the influence of adherence to growth hormone therapy with Norditropin® in children and teenagers in daily practice in Germany. This study will look mainly at the difference in near final height between children and teenagers who adhere to their therapy plan with Norditropin® to non-adherent patients. Participants will get Norditropin® as prescribed to them by their doctor. The study will last as long as the therapy with growth hormone is seen necessary by the participants' doctors and the participants, up to a maximum of 10 years. During the visits at the participants' doctors participants will be asked to fill in a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent of parent or legally acceptable representative of subject and child assent, as age-appropriate must be obtained before any study-related activities.

  1. The parent or legally acceptable representative of the child must sign and date the Informed Consent Form (according to local requirements) and
  2. The child must sign and date the Child Assent Form or provide oral assent (if required according to local requirements).
* The decision to initiate treatment with commercially available Norditropin® FlexPro® has been made by the treating physician and the patient's parents/legal guardian before and independently of the decision to include the patient in this study.
* Male or female, all age groups equal to or below 15 years with more than 2 years expected remaining treatment time until reaching NFH. Patients who self-inject should be above 8 years of age in order to be able to fill in the questionnaire.
* Children being GH naïve at baseline with one of the following confirmed diagnoses

  1. Isolated growth hormone deficiency (iGHD)
  2. Small for gestational age (SGA)

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* Patients who have an expected future duration of therapy of less than 2 years are not eligible for the study.

Ages: 0 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Paediatric patients with iGHD or SGA.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2019-06-21 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Near final height (NFH) standard deviation score (SDS) measured in scores | At the end of the study (up to 10 years)
  SDS, -3 to +3

SECONDARY OUTCOMES:
Change in growth rate (height velocity standard deviation score, HV SDS) | From baseline (month 0) to end of study (up to 10 years)
  Score, range -10 to +10
Change in growth rate (HV SDS) between visits (usually patients are seen every 3 to 6 months) | From baseline (month 0) to end of study (up to 10 years)
  Score, range -10 to +10
Adherence response as indicated in question at the bottom of newly developed Patient Reported Outcome (PRO) questionnaire each time questionnaire is filled out (preferably at each visit) | From baseline (month 0) to end of study (up to 10 years)
  The following adherence levels will be used:
  High adherence: above 85.7% of doses administered Medium adherence: 57.1 - 85.7% of doses administered Low adherence: below 57.1% of doses administered
Adherence measured as number of medication devices returned versus number of prescribed devices for the period between visits | From baseline (month 0) to end of study (up to 10 years)
  Count
Change of self-rated adherence level throughout the study measured in newly developed PRO questionnaire each time questionnaire is filled out (preferably at each visit) | From baseline (month 0) to end of study (up to 10 years)
  The following adherence levels will be used:
  High adherence: above 85.7% of doses administered Medium adherence: 57.1 - 85.7% of doses administered Low adherence: below 57.1% of doses administered

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Uniklinik Ulm - Dt. Zentrum für Kinder- und Jugendgesundheit (DZKJ), Ulm, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com